CLINICAL TRIAL: NCT05719805
Title: An Open-label, Randomized, Single-dose, 2-way Crossover Study to Establish Bioequivalence of 1 × 15-mg Mavacamten Capsule to 3 × 5-mg Mavacamten Capsules in Healthy Participants
Brief Title: A Study to Evaluate the Effects of Mavacamten in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CV027-1090
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Healthy Participants
Keywords: Hypertrophic cardiomyopathy (HCM); Left ventricular (LV) hypertrophy; Bioequivalence; Left Ventricular Outflow Tract Obstruction; Heart diseases; Cardiovascular diseases
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Hypertrophy; Ventricular Outflow Obstruction, Left; Heart Diseases; Cardiovascular Diseases | interventions — MYK-461

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mavacamten Dose 1 (Experimental)
  Interventions: Drug: Mavacamten
- Mavacamten Dose 2 (Experimental)
  Interventions: Drug: Mavacamten

INTERVENTIONS:
Drug: Mavacamten — Specified dose on specified days
  Other Names: MYK-461

SUMMARY:
The purpose of the study is to evaluate the effect between two different single doses of mavamten in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 32 kg/m^2, inclusive, at the screening visit.
* Healthy, as determined by physical examination, vital signs, 12-lead ECGs, and clinical laboratory assessments (including hematology, chemistry, and urinalysis) within the normal range at the screening visit and/or on Day -1. Participants with values outside of the normal range may be included if the values are not considered, by the investigator, to be clinically significant unless such values are explicitly excluded.
* Cytochrome P450 (CYP2C19) normal (*1/*1), rapid (*1/*17), or ultra-rapid (*17/*17) metabolizer, as determined by genotyping during screening.

Exclusion Criteria:

* Current or history of clinically significant cardiac condition, including but not limited to arrhythmia, LV systolic dysfunction, coronary heart disease; current, history, or family history of HCM; or evidence of prior myocardial infarction based on ECGs.
* Current or recent (within 3 months of study intervention administration) gastrointestinal disease including, but not limited to, bowel obstruction or perforation, gastrointestinal ulcers, esophageal varices, Crohn's disease, diverticulitis, irritable bowel syndrome, ileus, a gastrointestinal tract that is not anatomically intact, dyspepsia, constipation, diarrhea, or vomiting.
* Any gastrointestinal surgery (other than appendectomy) that, in the opinion of the investigator, could impact the absorption of study intervention.

Note: Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Predose and post-dose up to Day 80
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC [0-T]) | Predose and post-dose up to Day 80
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC [INF]) | Predose and post-dose up to Day 80

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) | Predose and post-dose up to Day 80
Terminal Half-life (T-Half) | Predose and post-dose up to Day 80
Number of Participants with Adverse Events (AEs) | Up to Day 80
Number of Participants with Serious AEs (SAEs) | Up to Day 80
Number of Participants with Vital Sign Abnormalities | Up to Day 80
Number of Participants with Electrocardiogram (ECG) Abnormalities | Up to Day 80
Number of Participants with Physical Examination Abnormalities | Up to Day 80
Number of Participants with Clinical Laboratory Abnormalities | Up to Day 80

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Local Institution - 0001, Miami, Florida
  - Local Institution - 0002, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome